CLINICAL TRIAL: NCT02970955
Title: Prospective Observational Study on a Risk Adaptive Scheme for Stereotactic Body Radiation Therapy (SBRT) for Medically Inoperable Thoracic Nodes Metastases
Brief Title: Prospecitve Observational Study on a Risk Adaptive Scheme for SBRT for Thoracic Nodes Metastases
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Medical Doctor, Istituto Clinico Humanitas
Other Study IDs: 1633
Record Dates: First submitted 2016-11-16; First posted 2016-11-22 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Thoracic Nodes Metastases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Inoperable thoracic nodes metastases: Oligometastatic patients with inoperable thoracic nodes metastases from any primary
  Interventions: Procedure: Inoperable thoracic nodes metastases

INTERVENTIONS:
Procedure: Inoperable thoracic nodes metastases — The radiation treatment will be delivered with three possible schedules, with a risk adaptive scheme according to number, site and size of metastatic nodes and based on the possibility to respect the constraints of healthy tissues

SUMMARY:
Oligometastatic patients with inoperable thoracic nodes metastases from any primary, except for hematologic malignancies, will undergo a risk adaptive scheme of stereotactic body radiation therapy (SBRT).

DETAILED DESCRIPTION:
The observational study is designed to evaluate safety and efficacy of a risk adaptive scheme of stereotactic body radiation therapy (SRT) in oligometastatic patients with thoracic nodes metastases, medically inoperable, using VMAT RapidArc approach. The potential advantage of this technique is the ability to deliver a more selective irradiation to tumour's target while reducing doses to normal tissue, optimizing the therapeutic window.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years with ECOG 0-2
* Karnofsky index > 70% (ECOG >2)
* Any primary, except for hematologic malignancies
* DFI (Disease-free interval) from diagnosis > 6 months
* Unresectable lesions or inoperable patients or patients who refused surgery
* Less than 3 metastatic thoracic nodes
* No extrathoracic disease or other metastatic sites stable or responding after chemotherapy, with less than 5 metastatic sites
* No life threatening conditions
* Chemotherapy completed at least 1 week before treatment
* Chemotherapy started at least 1 week after treatment allowed
* Systemic therapies other than chemotherapy allowed (i.e hormonal therapies and/or immunotherapy)
* Written informed consent

Exclusion Criteria:

* Previous RT in the same region
* Pregnant women
* Patients with inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inoperable thoracic nodes metastases from any primary, except for hematologic malignancies
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Local control of disease | 7 years
  Local control of the thoracic nodes stereotactic radiation therapy schedules for medically inoperable oligometastatic patients

SECONDARY OUTCOMES:
Progression-free survival for patients | 7 years
  A measure of the activity of the SBRT treatment on the disease by statistical methods
Overall survival for patients | 7 years
  Percentage of patients who are alive after a length of time
Quality of life evaluated by EORTC QLQ C30 questionnaires | 7 years
  At the end of the treatment and during the first follow-up appointment patients will complete the EORTC QLQ C30
Hematologic and non-hematologic toxicities | 7 years
  Hematologic and non-hematologic toxicities will be graded according to Common Terminology Criteria for Adverse Events version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Davide Franceschini, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Davide Franceschini, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franceschini D, Teriaca MA, Mancosu P, Bertolini A, Lo Faro L, Spoto R, Dominici L, Badalamenti M, Bellu L, Dei D, La Fauci F, Franzese C, Scorsetti M. Prospective phase II trial on ablative stereotactic body radiation therapy (SBRT) for medically inoperable thoracic nodes metastases. Radiother Oncol. 2024 Aug;197:110335. doi: 10.1016/j.radonc.2024.110335. Epub 2024 May 19. PMID 38772477